CLINICAL TRIAL: NCT05812430
Title: The Efficacy and Safety of Anlotinib Plus TQB2450 Combined With Nab-paclitaxel and Cisplatin as First-line Treatment for Advanced Biliary Tract Cancer
Brief Title: Anlotinib Plus TQB2450 Combined With Nab-paclitaxel and Cisplatin as First-line Treatment for Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hong Zong, Professor of Medicine, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-01
Record Dates: First submitted 2023-03-13; First posted 2023-04-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Advanced Biliary Tract Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib+TQB2450+nab-paclitaxel+cisplatin (Experimental)
  Interventions: Drug: anlotinib+TQB2450+nab-paclitaxel+cisplatin

INTERVENTIONS:
Drug: anlotinib+TQB2450+nab-paclitaxel+cisplatin — Anlotinib: 10mg, po, d1~14, q3w, until disease progression or unacceptable toxicity.
  TQB2450: 1200mg, ivgtt, d1, q3w, until disease progression or unacceptable toxicity.
  nab-paclitaxel: 200mg/㎡, ivgtt, d1, q3w, 6 cycles. cisplatin: 60mg/㎡, ivgtt, d1, q3w, 6 cycles.

SUMMARY:
To evaluate the efficacy and safety of anlotinib plus TQB2450 combined with nab-paclitaxel and cisplatin as first-line treatment for advanced biliary tract cancer

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-75 years old; both male and female are eligible.
* 2. Pathologically confirmed unresectable, untreated gallbladder cancer or intrahepatic/extrahapatic cholangiocarcinoma with at least one measurable lesion according to RECIST v1.1. Tissue samples must be provided for biomarker analysis, preferably newly acquired tissue. If newly acquired tissue is not available, 5-8 archived paraffin sections with a thickness of 5um must be provided.
* 3. ECOG score: 0-1.
* 4. Expected survival period ≥12 weeks.
* 5. Normal function of major organs, which meets the following criteria: Blood routine test: a) Hb ≥ 90 g/L (no blood transfusion within 14 days); b) ANC ≥ 1.5x 10^9/L; c) PLT ≥ 80x 10^9/L; Biochemical test: a) ALB ≥ 30g/L (no albumin transfusion within 14 days); b) ALT and AST <2.5ULN; if there is liver metastasis, ALT and AST ≤5ULN; c) TBIL ≤ 1.5ULN; d) plasma Cr ≤ 1.5ULN; or creatinine clearance rate (CCr) ≥60ml/min.
* 6. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%).
* 7. Participants must voluntarily agree to join the study, sign an informed consent form, and be able to comply with the visit and related procedures specified in the protocol. Female participants of childbearing potential or male participants whose partner is of childbearing potential must take effective contraceptive measures throughout the treatment period and for 6 months after the end of treatment.

Exclusion Criteria:

* 1. Confirmed allergy to anlotinib hydrochloride and/or its excipients, and TQB-2450 components;
* 2. Uncontrolled hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg), grade I or higher coronary heart disease, grade I arrhythmia (including QTc interval prolongation of >450 ms in males and >470 ms in females), and heart failure with urine protein positive;
* 3. Patients with clear gastrointestinal bleeding tendencies, including local active ulcer lesions and fecal occult blood (++), cannot be included. Patients with a history of black stool or vomiting within 2 months cannot be included;
* 4. Patients with abnormal coagulation function (INR > 1.5, APTT > 1.5 ULN) with a tendency to bleed;
* 5. Patients with multiple factors affecting oral drug absorption (such as dysphagia, nausea, vomiting, chronic diarrhea, and bowel obstruction, etc.);
* 6. Patients with central nervous system metastases;
* 7. Pregnant or lactating women;
* 8. Patients with other malignant tumors within 5 years (excluding cured skin basal cell carcinoma and cervical intraepithelial neoplasia);
* 9. Patients with a history of substance abuse that cannot be overcome or with mental illness;
* 10. Patients who participated in another drug clinical trial within 4 weeks;
* 11. Patients who have received VEGFR inhibitors such as sorafenib, sunitinib, or apatinib;
* 12. Patients with unhealed wounds or fractures;
* 13. Patients with abnormal thyroid function;
* 14. Urine protein ≥++ or 24-hour urine protein quantity greater than 1.0g;
* 15. Received target focus radiotherapy within 4 weeks prior to the first dose of study therapy;
* 16. Use of immunosuppressive drugs within 4 weeks prior to the first dose of study therapy, excluding nasal, inhalation or other routes of topical corticosteroids or physiological doses of systemic corticosteroids (i.e., not exceeding 10 mg/ day of prednisone or equivalent doses of other corticosteroids);
* 17. Receive live attenuated vaccine within 4 weeks before the first dose of study treatment or during the study period;
* 18. Had major surgical procedures (craniotomy, thoracotomy or laparotomy) or unhealed wounds, sores or fractures within 4 weeks prior to the first dose of study treatment;
* 19. Class 0 or 1 toxicity (excluding hair loss, non-clinically significant, and asymptomatic laboratory abnormalities) that did not return to National Cancer Institute General Adverse Event Terminology 4.03 (NCI CTCAE 4.03) due to prior antitumor therapy prior to the first dose of study therapy;
* 20. Symptomatic central nervous system metastases and/or cancerous meningitis are known. Subjects who had previously received BMS Eligible for study participation if BMS have remained stable for at least 4 weeks prior to the first dose of investigational therapy; And neurological symptoms must have returned to NCI CTCAE 4.03 level 0 or 1;
* 21. Active, known or suspected autoimmune disease or previous 2-year history of the disease (patients with vitiligo, psoriasis, alopecia, or Grave's disease that did not require systemic treatment within the last 2 years, hypothyroidism requiring only thyroid hormone replacement therapy, and type 1 diabetes requiring only insulin replacement therapy were included);
* 22. Uncontrolled co-morbidity includes, but is not limited to: HIV-infected persons (HIV-antibody positive). Severe infections that are active or poorly controlled clinically;
* 23. Symptomatic congestive heart failure (New York Heart Association Grade II-IV) or symptomatic or poorly controlled arrhythmias.
* 24. Uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg) even with standard treatment;
* 25. Any arterial thromboembolic event, including myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, occurred in the 6 months prior to admission for treatment;
* 26. Significant malnutrition, such as the need for intravenous nutritional solutions; Malnutrition corrected for more than 4 weeks prior to the first dose of study therapy was excluded;
* 27. A history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within the 3 months prior to enrollment (implantable port of intravenous infusion or catheter-derived thrombosis, or superficial venous thrombosis was not considered "severe" thromboembolism);
* 28. Uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or cancers that may lead to higher medical risk and/or uncertainty in the assessment of survival;
* 29. Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh grade B or more severe cirrhosis;
* 30. A history of ileus or the following: inflammatory bowel disease or extensive enterectomy (partial resection of the colon or extensive resection of the small intestine with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea;
* 31. Other acute or chronic diseases, psychiatric disorders, or abnormalities in laboratory test values that may increase the risk associated with study participation or study drug administration, or interfere with the interpretation of study results, and, in the investigator's judgment, classify patients as ineligible for study participation;
* 32. Known to have acute or chronic active hepatitis B (HBsAg positive with HBV DNA≥200 IU/mL or ≥103 copies /mL) or acute or chronic active hepatitis C (HCV antibody positive with HCV RNA positive);
* 33. A history of gastrointestinal perforation and/or fistula during the 6 months prior to study inclusion;
* 34. Suffers from interstitial lung disease;
* 35. Pregnant or nursing female patients;
* 36. Known history of primary immunodeficiency;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | about 2 years
  The RECIST1.1 standards were used to evaluate the efficacy of drugs.

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | about 2 years
Overall Survival(OS) | about 2 years
Disease Control Rate(DCR) | about 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: Undecided